CLINICAL TRIAL: NCT07122817
Title: Effects Of Emotional Suppression on Pain Perception and Physical Performance in Elderly Individuals
Brief Title: Emotional Suppression in Elderly Individuals
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Other Study IDs: 2025/231
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Elderly Person
Keywords: ELDERLY INDIVIDUALS; EMOTIONAL SUPPRESSION; PAIN PERCEPTION; PHYSICAL PERFORMANCE
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Individuals over 65 years of age who can independently carry out daily living activities and whose cognitive level is sufficient to understand and answer the surveys and tests in the study.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The group to be evaluated is comprised of individuals over 65 years of age, who can independently carry out their daily living activities, and whose cognitive level is sufficient to understand and answer the surveys and tests in the study.

SUMMARY:
The world's population is aging, and the proportion of individuals aged 60 and over is rapidly increasing. With aging, the prevalence of both physical and psychological health problems increases, negatively impacting quality of life. Chronic musculoskeletal pain, one of the most common health problems among older individuals, limits their daily activities and reduces their functional independence. Chronic pain is a complex experience that interacts not only with biological but also with psychological and social factors.

In this context, an individual's emotional regulation strategies play a crucial role in understanding the pain experience. Emotional suppression, in particular, is defined as the conscious suppression or inability to express one's emotions. This strategy has been reported to be associated with increased psychological stress, anxiety, depression, and pain sensitivity in the long term. Individuals who suppress their emotions have been shown to perceive pain as more threatening and develop more negative coping strategies.

Furthermore, cognitive tendencies such as pain catastrophizing, combined with emotional suppression, appear to increase an individual's psychological response to pain, impacting both pain intensity and psychological pain sensitivity. Such negative emotional regulation strategies can lead to increased pain perception and avoidance of physical activity, resulting in decreased physical performance.

Physical performance in older individuals is one of the key indicators determining their level of independence and quality of life. Tests such as the Timed Up and Go Test, the 6-Minute Walk Test, and the 30-Second Sit-to-Stand Test are widely used to assess mobility, balance, lower extremity endurance, and overall physical fitness. Chronic pain and its accompanying emotional factors are known to negatively impact physical performance.

However, studies examining the combined effects of emotional suppression on both pain perception and physical performance in older individuals are quite limited. This study contributes to the literature by offering a holistic assessment perspective by considering the physiological consequences of emotional regulation strategies in a multidimensional manner. Addressing the psychological and physical health of older individuals in conjunction is crucial for developing effective intervention programs. In this respect, the aim of the study was to examine the effect of the level of emotional suppression on pain perception (intensity and catastrophizing) and physical performance in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,
* Individuals who can independently carry out their daily living activities,
* Those with a cognitive level sufficient to understand and answer the surveys and tests in the study (Mini-Mental State Examination [MMSE] ≥ 24),
* Individuals who voluntarily agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Individuals with a history of serious neurological (e.g., stroke, Parkinson's disease, dementia), psychiatric (e.g., schizophrenia, bipolar disorder), or cardiopulmonary disease;
* Those with a history of acute injury, trauma, or surgery (within the last 6 months) that could affect pain perception or physical performance;
* Those who regularly use opioids or strong analgesic medications for pain;
* Individuals who are unable to complete assessment tests due to profound hearing or vision loss;
* Individuals diagnosed with severe depression and/or receiving active psychotherapy/psychiatric treatment;
* Individuals with physical or cognitive limitations that prevent them from completing surveys and performance tests.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Individuals over 65 years of age who can independently carry out daily living activities and whose cognitive level is sufficient to understand and answer the surveys and tests in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Scale | 4 weeks
  The Emotion Regulation Scale will be used in the study to assess participants' tendency to suppress their emotions. The Emotion Regulation Scale is a self-report scale developed by Gross and John that measures how individuals regulate their emotions. The Emotion Regulation Scale consists of two subscales: Cognitive Reappraisal and Expressive Suppression. Specifically, the emotional suppression subscale will be used in this study. Participants evaluate statements given to them on a 7-point Likert-type scale (1 = "Strongly disagree", 7 = "Strongly agree"). High scores on the scale indicate a high tendency to suppress emotional reactions. The Emotion Regulation Scale is a measurement tool widely used in psychological research with proven validity and reliability.
Pain Catastrophizing Scale | 4 weeks
  The Pain Catastrophizing Scale will be used to assess participants' cognitive and emotional responses to pain. The Pain Catastrophizing Scale, developed by Sullivan and colleagues, is a self-report scale that assesses negative thought patterns associated with pain. The scale consists of three subscales: Rumination, Magnification, and Helplessness, and a total of 13 items. Participants rate each item on a 5-point Likert-type scale, with "0 = Never" and "4 = Always." The total score ranges from 0 to 52, with higher scores indicating a greater psychological sensitivity to pain and a greater level of catastrophizing. The Pain Catastrophizing Scale is an effective tool for understanding the psychological factors that play a significant role in the subjective experience of pain, and its validity and reliability have been tested in various populations.
Numeric Pain Rating Scale | 4 weeks
  The Numeric Pain Rating Scale is a simple and common self-report tool used to assess participants' pain intensity. Participants are asked to rate their pain on a numerical scale from 0 (no pain) to 10 (unbearable pain). The Numeric Pain Rating Scale allows for quick and reliable measurement of subjective pain intensity and is widely used in clinical and research settings. The scale's validity and reliability have been demonstrated in several studies.
Brief Pain Inventory | 4 weeks
  The Brief Pain Inventory is a multidimensional pain measurement tool that assesses pain severity and its impact on activities of daily living. The scale collects information on pain severity (pain intensity), functional limitations caused by pain (emotional state, walking, sleep, etc.), and pain management methods. Participants rate pain on a scale of 0 (no pain) to 10 (worst pain). The Brief Pain Inventory is a highly valid and reliable tool for the clinical assessment of chronic pain and in research.
Timed Up and Go Test | 4 weeks
  The Timed Up and Go Test is a practical and valid performance test used to assess individuals' mobility, balance, and functional movement abilities. In the test, the participant rises from a chair, walks 3 meters, returns, and sits back down. Test duration is measured in seconds; shorter times indicate better functional performance. The Timed Up and Go Test is widely used to identify fall risk and mobility limitations, particularly in older individuals.
Chair Stand Test | 4 weeks
  Chair Stand Test will be used to measure lower body strength, which is important for everyday activities like climbing stairs and getting up from a chair. The participant sits in the middle of a chair with arms crossed at the wrists and held against the chest. On the command "Go," the participant stands up fully and then sits back down as many times as possible within 30 seconds.The number of full stands completed reflects lower body strength and endurance, which are crucial for maintaining independence and mobility.
Arm Curl Test | 4 weeks
  Arm Curl Test will be used to evaluate upper body strength, particularly the strength of the biceps, which is important for lifting and carrying objects.The participant sits on a chair, holding a dumbbell (usually 5 lbs for women, 8 lbs for men) in the dominant hand with the arm fully extended. The participant curls the arm by bending the elbow and bringing the dumbbell up to shoulder height, then lowers it back down. The test lasts 30 seconds, counting the number of curls completed. The total number of curls completed shows upper body strength endurance, necessary for daily tasks like carrying groceries.
Chair Sit-and-Reach Test | 4 weeks
  Chair Sit-and-Reach Test will be used to assess the flexibility of the lower body, especially the hamstrings and lower back, which affect posture and movement.The participant sits on the edge of a chair and extends one leg straight out with the heel on the floor and toes pointing upward. Keeping the back straight, the participant reaches forward toward the toes as far as possible without bouncing.
  The distance (measured in inches or centimeters) reached beyond the toes (positive if past toes, negative if not reaching toes) reflects lower body flexibility, important for safe mobility and fall prevention.
Back Scratch Test | 4 weeks
  Back Scratch Test will be used evaluate upper body (shoulder) flexibility, which affects activities like reaching overhead or behind the back. The participant reaches one hand over the shoulder and down the back, while the other hand reaches up the middle of the back from the waist. The goal is to touch or overlap the middle fingers of both hands. The distance between the fingertips is measured. The gap or overlap between fingers (measured in inches or centimeters) reflects shoulder flexibility, essential for daily tasks like grooming or dressing.
Foot Up-and-Go Test | 4 weeks
  Foot Up-and-Go Test will be used to assess agility, balance, and speed of movement, which are critical for preventing falls and moving safely. Starting seated in a chair, the participant stands up, walks 8 feet (2.44 meters), turns around, and returns to the chair as quickly as possible without running. The time taken to complete the task is recorded. The total time reflects the participant's agility and dynamic balance; shorter times indicate better functional mobility.
6-Minute Walk Test | 4 weeks
  6-Minute Walk Test wil be used to measure aerobic endurance, which is important for stamina in daily activities like walking or climbing stairs.
  Procedure:
  The participant walks back and forth along a marked walkway (usually 50 feet or 15 meters) for 6 minutes at a comfortable, steady pace. The total distance covered in 6 minutes is recorded.
  What it indicates:
  The distance walked indicates cardiovascular fitness and endurance; longer distances mean better aerobic capacity.

SECONDARY OUTCOMES:
Geriatric Depression Scale: | 4 weeks
  The Geriatric Depression Scale is a self-report-based screening tool developed to detect symptoms of depression in older adults. The scale is available in two versions: short and long; the 15-item short form was used in our study. The items consist of simple statements answered with "Yes" or "No" and assess the presence of depressive symptoms. The Geriatric Depression Scale has high reliability and validity in the elderly population and is widely used in research as well as in clinical/practice settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided